CLINICAL TRIAL: NCT04030728
Title: A Randomized, Controlled Study of Standardized Patient Coaching Versus Patient Management According to Local Practice for Patients With Hormone Receptor Positive HER2 Negative Metastatic Breast Cancer Treated With Abemaciclib
Brief Title: Implementing Patients´ Competence in Oral Breast Cancer Therapy
Acronym: IMPACT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Onco Medical Consult GmbH (Industry)
Collaborators: Eli Lilly and Company (Industry); Institut fuer Frauengesundheit (Other)
Responsible Party: Sponsor
Other Study IDs: OMC2018/01
Record Dates: First submitted 2019-07-04; First posted 2019-07-24 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer
Keywords: patient coaching; Advanced or metastatic breast cancer; Abemaciclib; hormone receptor positive (HR+); human epidermal growth factor receptor 2 (HER2) negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Standardized coaching arm: Patients in this group receive a continuous standardized MOATT based patient education and coaching and optional eMBSR (electronic Mindfulness-Based Stress Reduction) within the first 24 weeks of Abemaciclib treatment.
- Group 2: Coaching according to local practice: Patients in this group receive a patient management according local routine.

SUMMARY:
The aim of the IMPACT - Implementing Patients' competence in oral breast cancer therapy - study is to evaluate the effectiveness of a standardized patient education and coaching and optional eMBSR for therapy management provided by specially trained oncology nurses regarding persistence rate, side effects management and unplanned therapy interruptions in outpatient oncology care for patients under Abemaciclib treatment.

DETAILED DESCRIPTION:
Breast cancer therapy has advanced by far over the last decade. Introduction of novel therapies as well as the introduction of mammography screening are thought to have reduced mortality over the last decade. More women are treated on an individual basis, trying to avoid toxic and non-effective therapies.

However, every year about 18.000 women are diagnosed with metastastic breast cancer in Germany. Breast cancer remains one of the main reasons for deaths among women and is the main reason for death due to cancer in younger women.

Once a tumor is metastasized, well balanced treatment decisions have to be made to take both into consideration, a high chance of tumor control and a low risk for side effects. Especially in the metastatic setting symptom control and quality of life need to be in the focus of the therapy and patient care.

Modern anticancer strategies are designed against specific molecular targets with the goal of sparing normal, non-neoplastic tissues. Choosing specific molecular targets, however, is problematic. CDK4/6 (Cyclin dependent kinase 4 and 6) are important candidate targets for therapeutic intervention.

Traditionally, anticancer therapy has been dominated by intravenous drug therapy. However, oral agents, like CDK4/6 inhibitors, provide an attractive approach to this kind of treatment and use of oral treatments is increasing. Currently, there are three CDK4/6 inhibitors that have reached clinical practice in the management of ER+ HER2- advanced disease. One of them is Ademaciclib which is approved in the US since September 2017 for "adult patients who have hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative advanced or metastatic breast cancer that has progressed after taking therapy that alters a patient's hormones".

Oral agents for cancer treatment are increasingly prescribed due to their benefits. However, this type of therapy requires a high level of self-management competence by the patient. A standardized patient education provided by physicians and oncology nurses may influence the handling of the oral agents in a positive way regarding side effects and unplanned therapy interruptions.

When it comes to oral agents, the place of treatment is the patients' home. In this treatment setting, correct treatment management cannot be utilized without identifying a patient's needs to be empowered to become an expert of his/her treatment because cancer therapies are commonly difficult to handle and the medication often shows a high risk of side effects and interactions with other drugs. Care providers are challenged by the question of how mostly elderly and multimorbid patients and their supporting relatives can be enabled with essential competencies to manage their treatment by themselves. Before patients start their cancer therapy, they are usually provided with information about the treatment by their physician. However, patients often feel overwhelmed by all the details in this stressful situation and tend to have a reduced capacity to assimilate complex information. Education and additional support at the beginning and in the course of the treatment can be a useful approach for patients to better handle this situation.

Recent studies showed the positive impact of supportive care programs on patients provided by nurses. Patient-focused motivation techniques and education performed by nurses are suitable to strengthen the patients' understanding of risks and benefits from the anti-cancer treatment and oral agents. These care programs can prevent an incorrect medication intake due to misunderstandings, lead to a decrease of treatment-related symptoms like pain and fatigue and reduce critical events. In addition, patient education can facilitate supportive care through a better communication between patient and health care provider and may advance the early detection of adverse toxicity events and foster rapid symptom management.

Mindfulness based stress reduction (MBSR) shows a positive effect on mental health in breast cancer patients. The evidence confirms that MBSR reduces anxiety, depressiveness and stress of breast cancer patients and increases the health-related quality of life. A key ingredient to reduce the damaging effects of chronic stress, reducing distress, and improving quality of life is to have patients engage in behaviors that decrease sympathetic and increase parasympathetic arousal. Studies show that MBSR have a positive effect on many systems in our body and create fundamental changes in the way the brain functions. MBSR can affect neurotransmitters (i.e. glutamate, GABA) and neuromodulators (i.e. dopamine, serotonin, epinephrine), which are essential in maintaining a healthy balance between sympathetic and parasympathetic arousal, therefore, helping to manage the stress response.

The aim of the IMPACT - Implementing Patients' competence in oral breast cancer therapy - study is to evaluate the effectiveness of a standardized patient education and coaching and optional eMBSR for therapy management provided by specially trained oncology nurses regarding persistence rate, side effects management and unplanned therapy interruptions in outpatient oncology care for patients under Abemaciclib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult breast cancer patients (age ≥18 years).
* Patients with HR+, HER2- advanced or metastatic breast cancer proven by clinical measures (i. e. standard imaging) whose disease has progressed after hormonal therapy in combination with fulvestrant, or alone in women whose disease has progressed after hormone therapy and prior chemotherapy (advanced disease must not be amenable to resection with curative intent).
* Patients treated with Abemaciclib according to the SmPC and each center´s medical practice.
* Informed consent prior to onset of documentation.

Exclusion Criteria:

* Patients with serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Females who are pregnant or lactating.
* Patients with active bacterial infections (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infections, or detectable viral infections (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
* Patients with a personal history in the past 5 years of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Patients with contraindications against Abemaciclib according to respective SmPC´s.
* Patients who are not eligible for observation due to severe comorbidities other then mentioned above or unavailability according to the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffer from HR+, HER2- advanced or metastatic breast cancer treated with with orally administered commercially available, prescribed Abemaciclib in combination with an aromase inhibitor or fulvestrant as initial endocrine-based therapy or in women who have received prior endocrine therapy, thereby reflecting the current SmPC (Fachinformation Verzenios®). All treatments are prescribed and performed according to each center's medical practice. Any treatment choice or change in regimen is performed at the discretion of each treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
(Potential) difference in persistence rate after 24 weeks of Abemaciclib therapy in both study arms. | 24 weeks
  The primary objective of this study is to evaluate both study arms regarding the (potential) effect of patient management according to local routine versus continuous standardized patient education and coaching using the MOATT on persistence rate within the first 24 weeks of Abemaciclib treatment.

SECONDARY OUTCOMES:
Patient decided interruptions | 24 weeks
  Total time of patient decided interruptions in days during 24 weeks of Abemaciclib therapy in both study arms.
eMSBR | 24 weeks
  The effect of eMSBR after 24 weeks of Abemaciclib therapy.
Quality of life assessed by the FACT-B (Version 4.0) questionnaires. | 24 weeks
  After weeks 2, 6, 12, 18 and 24, quality of Life (QoL) will be assessed by the FACT-B (Version 4.0) questionnaires.
Patient distress assessed via distress thermometer. | 24 weeks
  After weeks 2, 6, 12, 18 and 24, patient distress will be assessed via distress thermometer.
To assess patient reported self-efficacy: patient diary | 24 weeks
  Self-efficacy will be patient reported and surveyed through a patient dairy.
To assess patient reported side-effects. | 24 weeks
  Type and duration of side-effects will be patient reported and surveyed through a patient dairy.
To assess patient reported health related stress. | 24 weeks
  Health related stress will be patient reported and surveyed via distress thermometer questionnaire.
To assess patient reported therapy related knowledge. | 24 weeks
  Therapy related knowledge will be surveyed via MOATT (MASCC Oral Agent Teaching Tool).
Incidence of therapy interruptions. | 24 weeks
  Amount of relevant events will be surveyed through patient self-reporting via patient diary.
Duration of therapy interruptions. | 24 weeks
  Relevant events (in days) will be surveyed through patient self-reporting via patient diary.
Safety and tolerability of Abemaciclib treatment: NCI Common Toxicity Criteria Version 5.0 | 24 weeks
  Incidence of adverse events and serious adverse events will be reported according to NCI Common Toxicity Criteria Version 5.0.
Efficacy between the two study arms at week 24 in routine clinical practice as assessed by Progression free survival rate (PFS). | 24 weeks
  Progression free survival (PFS) rate at 24 weeks of therapy. PFS is defined as time interval from start of therapy until progressive proven with clinical measures according to expertise and daily clinical routine or death from any cause, whichever comes first.
Efficacy between the two study arms at week 24 in routine clinical practice as assessed by Overall survival rate (OS). | 24 weeks
  Overall survival (OS) rate at 24 months is defined as the time to death from therapy start of Abemaciclib.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Tesch, Prof. Dr. med., Principal Investigator — Onkologie Bethanien Frankfurt; Manfred Welslau, Dr. med., Principal Investigator — Onkologie Aschaffenburg

REFERENCES:
- [Background] Bock K, Heywang-Kobrunner S, Regitz-Jedermann L, Hecht G, Kaab-Sanyal V. [Mammography screening in Germany. Current results and future challenges]. Radiologe. 2014 Mar;54(3):205-10. doi: 10.1007/s00117-013-2581-7. German. PMID 24623009
- [Background] Eisemann N, Waldmann A, Katalinic A. Epidemiology of Breast Cancer - Current Figures and Trends. Geburtshilfe Frauenheilkd. 2013 Feb;73(2):130-135. doi: 10.1055/s-0032-1328075. PMID 24771909
- [Background] Kolberg HC, Luftner D, Lux MP, Maass N, Schutz F, Fasching PA, Fehm T, Janni W, Kummel S. Breast Cancer 2012 - New Aspects. Geburtshilfe Frauenheilkd. 2012 Jul;72(7):602-615. doi: 10.1055/s-0032-1315131. PMID 25324576
- [Background] Maass N, Schutz F, Fasching PA, Fehm T, Janni W, Kummel S, Kolberg HC, Luftner D, Wallwiener M, Lux MP. Breast Cancer Update 2014 - Focus on the Patient and the Tumour. Geburtshilfe Frauenheilkd. 2015 Feb;75(2):170-182. doi: 10.1055/s-0035-1545704. PMID 25797960
- [Background] Loehberg CR, Almstedt K, Jud SM, Haeberle L, Fasching PA, Hack CC, Lux MP, Thiel FC, Schrauder MG, Brunner M, Bayer CM, Hein A, Heusinger K, Heimrich J, Bani MR, Renner SP, Hartmann A, Beckmann MW, Wachter DL. Prognostic relevance of Ki-67 in the primary tumor for survival after a diagnosis of distant metastasis. Breast Cancer Res Treat. 2013 Apr;138(3):899-908. doi: 10.1007/s10549-013-2460-y. Epub 2013 Mar 12. PMID 23479421
- [Background] Fasching PA, Brucker SY, Fehm TN, Overkamp F, Janni W, Wallwiener M, Hadji P, Belleville E, Haberle L, Taran FA, Luftner D, Lux MP, Ettl J, Muller V, Tesch H, Wallwiener D, Schneeweiss A. Biomarkers in Patients with Metastatic Breast Cancer and the PRAEGNANT Study Network. Geburtshilfe Frauenheilkd. 2015 Jan;75(1):41-50. doi: 10.1055/s-0034-1396215. PMID 25684786
- [Background] Wadler S. Perspectives for cancer therapies with cdk2 inhibitors. Drug Resist Updat. 2001 Dec;4(6):347-67. doi: 10.1054/drup.2001.0224. PMID 12030783
- [Background] Banna GL, Collova E, Gebbia V, Lipari H, Giuffrida P, Cavallaro S, Condorelli R, Buscarino C, Tralongo P, Ferrau F. Anticancer oral therapy: emerging related issues. Cancer Treat Rev. 2010 Dec;36(8):595-605. doi: 10.1016/j.ctrv.2010.04.005. Epub 2010 Jun 8. PMID 20570443
- [Background] Schilder CM, Seynaeve C, Linn SC, Boogerd W, Beex LV, Gundy CM, Nortier JW, van de Velde CJ, van Dam FS, Schagen SB. Cognitive functioning of postmenopausal breast cancer patients before adjuvant systemic therapy, and its association with medical and psychological factors. Crit Rev Oncol Hematol. 2010 Nov;76(2):133-41. doi: 10.1016/j.critrevonc.2009.11.001. Epub 2009 Dec 24. PMID 20036141
- [Background] May P, Figgins B. Oral anticancer therapy: a comprehensive assessment of patient perceptions and challenges. J Community Support Oncol. 2016 Mar;14(3):112-6. doi: 10.12788/jcso.0226. PMID 27058868
- [Background] Molassiotis A, Brearley S, Saunders M, Craven O, Wardley A, Farrell C, Swindell R, Todd C, Luker K. Effectiveness of a home care nursing program in the symptom management of patients with colorectal and breast cancer receiving oral chemotherapy: a randomized, controlled trial. J Clin Oncol. 2009 Dec 20;27(36):6191-8. doi: 10.1200/JCO.2008.20.6755. Epub 2009 Nov 16. PMID 19917849
- [Background] Bordonaro S, Romano F, Lanteri E, Cappuccio F, Indorato R, Butera A, D'Angelo A, Ferrau F, Tralongo P. Effect of a structured, active, home-based cancer-treatment program for the management of patients on oral chemotherapy. Patient Prefer Adherence. 2014 Jun 25;8:917-23. doi: 10.2147/PPA.S62666. eCollection 2014. PMID 25028540
- [Background] Chau I, Legge S, Fumoleau P. The vital role of education and information in patients receiving capecitabine (Xeloda). Eur J Oncol Nurs. 2004;8 Suppl 1:S41-53. doi: 10.1016/j.ejon.2004.06.008. PMID 15341881
- [Background] Temel JS, Greer JA, Admane S, Gallagher ER, Jackson VA, Lynch TJ, Lennes IT, Dahlin CM, Pirl WF. Longitudinal perceptions of prognosis and goals of therapy in patients with metastatic non-small-cell lung cancer: results of a randomized study of early palliative care. J Clin Oncol. 2011 Jun 10;29(17):2319-26. doi: 10.1200/JCO.2010.32.4459. Epub 2011 May 9. PMID 21555700
- [Background] Campbell CP. An oral cancer therapy nurse navigator role. Can Nurse. 2016 Apr;112(3):26-7. No abstract available. PMID 27373026
- [Background] Cramer H, Lauche R, Paul A, Dobos G. Mindfulness-based stress reduction for breast cancer-a systematic review and meta-analysis. Curr Oncol. 2012 Oct;19(5):e343-52. doi: 10.3747/co.19.1016. PMID 23144582
- [Background] Chaoul A, Milbury K, Sood AK, Prinsloo S, Cohen L. Mind-body practices in cancer care. Curr Oncol Rep. 2014 Dec;16(12):417. doi: 10.1007/s11912-014-0417-x. PMID 25325936
- [Background] Carlson LE, Doll R, Stephen J, Faris P, Tamagawa R, Drysdale E, Speca M. Randomized controlled trial of Mindfulness-based cancer recovery versus supportive expressive group therapy for distressed survivors of breast cancer. J Clin Oncol. 2013 Sep 1;31(25):3119-26. doi: 10.1200/JCO.2012.47.5210. Epub 2013 Aug 5. PMID 23918953
- [Background] Holzel BK, Carmody J, Vangel M, Congleton C, Yerramsetti SM, Gard T, Lazar SW. Mindfulness practice leads to increases in regional brain gray matter density. Psychiatry Res. 2011 Jan 30;191(1):36-43. doi: 10.1016/j.pscychresns.2010.08.006. Epub 2010 Nov 10. PMID 21071182
- [Background] Matchim Y, Armer JM, Stewart BR. Mindfulness-based stress reduction among breast cancer survivors: a literature review and discussion. Oncol Nurs Forum. 2011 Mar;38(2):E61-71. doi: 10.1188/11.ONF.E61-E71. PMID 21356643
- [Background] Musial F, Bussing A, Heusser P, Choi KE, Ostermann T. Mindfulness-based stress reduction for integrative cancer care: a summary of evidence. Forsch Komplementmed. 2011;18(4):192-202. doi: 10.1159/000330714. Epub 2011 Aug 8. PMID 21934319
- [Background] Piet J, Wurtzen H, Zachariae R. The effect of mindfulness-based therapy on symptoms of anxiety and depression in adult cancer patients and survivors: a systematic review and meta-analysis. J Consult Clin Psychol. 2012 Dec;80(6):1007-20. doi: 10.1037/a0028329. Epub 2012 May 7. PMID 22563637
- [Background] Zainal NZ, Booth S, Huppert FA. The efficacy of mindfulness-based stress reduction on mental health of breast cancer patients: a meta-analysis. Psychooncology. 2013 Jul;22(7):1457-65. doi: 10.1002/pon.3171. Epub 2012 Sep 7. PMID 22961994
- [Background] Wurtzen H, Dalton SO, Elsass P, Sumbundu AD, Steding-Jensen M, Karlsen RV, Andersen KK, Flyger HL, Pedersen AE, Johansen C. Mindfulness significantly reduces self-reported levels of anxiety and depression: results of a randomised controlled trial among 336 Danish women treated for stage I-III breast cancer. Eur J Cancer. 2013 Apr;49(6):1365-73. doi: 10.1016/j.ejca.2012.10.030. Epub 2012 Dec 19. PMID 23265707
- [Background] Shennan C, Payne S, Fenlon D. What is the evidence for the use of mindfulness-based interventions in cancer care? A review. Psychooncology. 2011 Jul;20(7):681-97. doi: 10.1002/pon.1819. Epub 2010 Aug 4. PMID 20690112